CLINICAL TRIAL: NCT00561899
Title: Comparison of Safety, Tolerability and Efficacy of Three Drug Combinations for Intermittent Preventive Treatment in Children Aged 1-5 Years in an Area of Seasonal Malaria Transmission in Upper River Division, The Gambia
Brief Title: Comparison of Three Drug Combinations for Intermittent Treatment of Malaria in Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Department of State for Health and Social Welfare, The Gambia (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SCC1089; GMP_PII_6
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: safety; tolerability; efficacy; intermittent prevetive treatment; children
MeSH Terms: conditions — Malaria | interventions — Amodiaquine; piperaquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): SP+AQ
  Interventions: Drug: SP, amodiaquine, piperaquine, dihdroartemisinin
- 2 (Experimental): Piperaquine plus SP arm
  Interventions: Drug: intermittent preventive treatment
- 3 (Experimental): Du-Cotecxin
  Interventions: Drug: Du-Cotecxin

INTERVENTIONS:
Drug: SP, amodiaquine, piperaquine, dihdroartemisinin — once every month during september, October and November
  Other Names: Fansidar; Du-Cotecxin
  Arms: 1
Drug: intermittent preventive treatment — SP(500mg sulfadoxine/25mg pyrimethamine)1.25mg SP per kg stat Amodiaquine (200mg base) 25mg/kg over 3 days Piperaquine (320 mg per tablet) 16.8 g/kg daily for 3 days Du-Cotecxin ( 40mg dihydroartemisinin(DHA)/320mg piperaquine(PQP))PQP/DHA 1.6/12.8mg/kg once daily for 3 days
  Other Names: SP; Du-Cotecxin
  Arms: 2
Drug: Du-Cotecxin — Du-Cotecxin (40mg dihydroartemisinin (DHA/320mg Piperaquine (PQP) PQP/DHA 1.6/12.8mg/kg once daily for 3 days
  Other Names: SP
  Arms: 3

SUMMARY:
Intermittent preventive treatment (IPT) offers a way of preventing malaria infection without compromising the development of malaria immunity or encouraging drug resistance. The effect of IPT in children in the prevention of malaria has been evaluated in a number of trials in areas of seasonal malaria transmission. Results from these trials have shown that IPTc provided between 40% - 86% protection against clinical malaria. In 2006, a trial that compared two methods of IPTc delivery was carried out in Upper River Division, The Gambia. Preliminary results of the trial have shown that the treatment was very effective as only 4% (45/1133) of the children seen at the end of year cross-sectional survey were parasitaemic. Tolerability was assessed in a subset of 1100 children and the results showed that about 13.5% of children developed mild to moderate vomiting. Malaise was present in about 10% of the study subjects. Severe adverse events were rare. Thus it is important to investigate if other drug regimens might be equally effective in preventing malaria but less likely to cause adverse events. During the 2007 malaria transmission season, 1009 children aged 1-5 years will be individually randomized to receive amodiaquine plus SP, piperaquine plus SP or Artekin TM (dihdroartemisinin plus piperaquine) at monthly intervals on three occasions during the months of September, October, and November. To determine the prevalence of side effects following drug administration participants in each treatment group will be visited at home three and seven days after each round of drug administration and a side effects questionnaire completed. To help establish whether these adverse events are drug related, the same questionnaire will be administered after each treatment round, to 286 age-matched children who are not part of the trial. The primary ends points will be the incidence of adverse events.

DETAILED DESCRIPTION:
Objectives

Primary Objective To determine the safety and tolerability of amodiaquine(AQ) (three days) plus sulfadoxine-pyrimethamine(SP) (one day), piperaquine(PQP) (three days) plus SP (one day), and Artekin TM (PQP plus dihydroartemisinin, DHA) (3 days) when used for seasonal IPT in children.

Secondary Objective To determine the efficacy of AQ (three days) plus SP (one day), PQP (three days) plus SP (one day) and Artekin TM (3 days) when used for seasonal IPT in children.

3.4 Randomisation Open-label, individual randomisation was carried out three weeks before the first dose of IPTc administration in September 2007. Study subjects were individually randomised into either the AQ plus SP, PQP plus SP or ArtekinTM treatment groups in a 1:1:1 fashion. An independent statistician generated the randomizing subject study number (SSN) that assigned each SSN to one of the treatment groups. A photo ID card was given to all participants to facilitate identification at every contact, at home or in the health centres.

3.5 Drug distribution at the health centres Study subjects and their parents were informed about the date of treatment approximately one week before any intervention. Treatment is scheduled to be given during the months of September, October and November. Drugs are to be given at the nearest health centre by a designated member of staff. Tablets are crushed, mixed with honey or suspended in water and given on a spoon. Staff who administer drugs at the health centre play no further part in the trial. All participants are kept under observation for 30 minutes after drugs are taken. In case of vomiting, the drug is re-administrated. At the time of each monthly drug administration, a brief clinical assessment is carried out. Children who are febrile are screened for malaria using a rapid antigen test. Children found to have malaria are treated with Lumefantrine-artemether (CoartemTM, Norvatis Pharma., Basel Switzerland).

3.7 Morbidity surveillance during the rainy season Passive surveillance for malaria will be maintained throughout the transmission season. Parents/guardians are being encouraged to take their children to the health centre identified as being closest to their home at any time that their child becomes unwell. Project staff are based at each of these health facilities to identify children in the trial and to ensure that they are seen, properly investigated and treated promptly. At each clinic visit, axillary temperature is recorded using a digital thermometer and haemoglobin concentration measured using a Hemocue machine. A dipstick for diagnosis of malaria is to be used if fever (axillary temperature of ³ 37.5°C) or a history of fever within the previous 48 hours is present. In such cases, a thick blood smear is also be collected for subsequent confirmation of the diagnosis. Study subjects with documented fever (axillary temperature of ³ 37.5°C) or history of recent fever and malaria parasitaemia are treated with Coartem. The treatment of study subjects seen at the health centres for other conditions is being carried out in accordance with national guidelines.

3.8 End of malaria transmission season cross-sectional survey Children enrolled in the study will be seen at the OPD clinic at the end of malaria transmission season for examination by a study physician and a finger-prick blood sample will be obtained for preparation of a thick blood smear and determination of haemoglobin concentration. A standardized questionnaire will be administered to the parents/guardians of the study subject, to collect information regarding illness that had occurred since the last visit, symptoms experienced, use of healthcare facilities and use of medicines. Information on the use of bed nets will be collected again at this visit.

3.10. Assessment of adverse events To determine the prevalence of minor side effects following drug administration such as headache, fever, weakness, abdominal pain, anorexia, nausea, vomiting, diarrhoea, rash, itching or sleep disorder participants in each treatment group are to be visited at home three and seven days after each round of drug administration and a side effects questionnaire completed. Field workers who complete these questionnaires will be unaware of the treatment group to which the child belongs. To help establish whether these adverse events are drug related, the same questionnaire will be administered once after each treatment round, to 286 children who are not part of the trial, recruited from nearby villages and matched for age to children in the trial.

Any serious adverse event that occurs during the study period will be reported to the Local Safety Monitor and Chairman of DSMB.

Primary end-point:

- Incidence of any adverse events during the observation period.

Secondary endpoints:

* Mean Hb (g/dl) at the end of malaria transmission.
* Prevalence of malaria parasitaemia at the end of the malaria transmission season.
* Number of OPD attendances with malaria that meet the case definitions as indicated below during the surveillance period.

Data management and analysis All baseline, surveillance and laboratory data will be collected on forms designed for the trial. Field and laboratory staff will be trained to follow the procedures set out in a series of Standard Operating Procedures (SOPs). Key data will be double entered and inconsistencies checked; range checks will be used for standard variables. Primary analyses will be performed on an intention to treat (ITT) basis. Any child who receives a first dose of drug will be included in the ITT analysis. Children who are randomised but who do not receive any mediation will not be included in this analysis.

Sample size calculations Drugs for IPT need to be acceptable and have low frequency of adverse events. If the frequency of adverse events is 20% in the SP/AQ group, a trial with 286 children per arm has 90% power to detect a halving in the frequency of adverse events, using a significance level of 0.05, or a reduction to 9% or less if a significance of 0.025 is used (to preserve an overall type 1 error rate of 5% for the primary endpoint when there are 2 comparisons, each alternative drug group with SP/AQ). If the frequency of adverse events is 15%, a reduction to 5% or less can be detected with the same power, and if the frequency is 10% a reduction to 2% or less can be detected. Based on experience from several studies the drop-out rate is not expected to exceed 15% and is likely to be less. Allowing for 15% drop out, a sample size of 286*3/(1-0.15)=1009 is needed.

Withdrawal during the study:

Study subjects may be withdrawn from the study for any one of the following reasons.

1. Withdrawal of parental / legal guardian's consent.
2. Serious adverse event attributable to the study drug.
3. Loss to follow-up.

Children who develop adverse events attributable to study drugs should not receive further doses but should be followed-up to monitor safety until the resolution of the adverse reaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 1 to 5 years at enrolment.
2. Informed consent obtained from parents or legal guardians.
3. No current participation in another malaria intervention trial.
4. Free of obvious health problems as established by medical history and clinical examination before entering into the study.
5. Available for the duration of the study.

Exclusion Criteria:

1. Known allergy to any of the antimalarial drugs used in the trial and if this is unknown, then a history of allergic reaction to any drug.
2. Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory tests.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1295 (Actual)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of AQ plus SP, PQP plus SP, and PQP plus DHA when used for seasonal IPT in children | Onset of IPT to end of malaria season

SECONDARY OUTCOMES:
The efficacy of the three drug regimens when used for seasonal IPT in children | Onset of IPT to end of malaria season

CONTACTS AND LOCATIONS:
Overall Officials: Kalifa Bojang, MD, Principal Investigator — Medical Research Council Unit, The Gambia; Kalifa Bojang, MD, Principal Investigator — Medical Research Council
Locations (1):
- Medical Research Council Laboratories,, Banjul, The Gambia

REFERENCES:
- [Derived] Bojang K, Akor F, Bittaye O, Conway D, Bottomley C, Milligan P, Greenwood B. A randomised trial to compare the safety, tolerability and efficacy of three drug combinations for intermittent preventive treatment in children. PLoS One. 2010 Jun 21;5(6):e11225. doi: 10.1371/journal.pone.0011225. PMID 20574538